CLINICAL TRIAL: NCT05110755
Title: Correlation of Physical Activity and Respiratory Health in COPD Patient
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/Lhr/0319 Misdaq Batool
Record Dates: First submitted 2021-08-17; First posted 2021-11-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Respiratory Health; Pulmonary Function; Physical Activity; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COPD is a common, preventable and treatable disease that is characterized by persistent respiratory symptoms and airflow limitation that is due to airway and/or alveolar abnormalities, usually caused by significant exposure to noxious particles or gases. COPD is third leading cause of death worldwide. "Ideal cardiovascular health," a set of factors, including several directly along the causal pathway of transitions from health to disease, that protect against the development of cardiac disease. Working definition of respiratory health are the dual concepts of pulmonary reserve, as reflected by peak lung function in young adulthood, and susceptibility, as reflected by risk for future accelerated decline in lung function after the attainment of this peak. There is relationship between physical activity, disease severity, health status and prognosis in patients with COPD. Common pulmonary function tests include spirometry, lung volumes, and diffusing capacity for carbon monoxide (DLCO). Spirometry assesses airflow limitation. Diffusing capacity for carbon monoxide provides information on the health of alveolar-capillary membrane.

This study will be cross-sectional correlational study. It will find correlation between person's physical activity and respiratory health. IPAQ and 6MIN walk test will be used as measuring tools of physical activity and FEV1 and TLV for estimating respiratory health. Spirometer will be used to measure respiratory health. Data will be collected from different hospital settings and analysed using SPSS software. All ethical considerations will be followed.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a heterogeneous and multisystemic disease with progressive increasing morbidity and mortality. Chronic obstructive pulmonary disease (COPD) is a deteriorating respiratory disease with some extrapulmonary effects that contribute to disease severity in patient. The etiology, in general, involves exposure to external noxious particles or gases. In the Western world this is particularly a result of (cigarette) smoking and in the non-Western world it is mainly a result of indoor cooking. COPD pathology is driven by chronic inflammation, which continues to be observed after stopping smoking, even after ⩾1 year. The combination of the exposure and inflammation leads to lung tissue damage, resulting in remodeling of the lung.Global Burden of Disease programme in 2010 identified chronic obstructive pulmonary disease (COPD) as the third leading cause of death worldwide up from 4th in 1990. This high mortality due to COPD is caused due to smoking and rapidly aging population. China alone contributed to about one-third (0.9million/year) of all deaths from COPD worldwide. Within China, the prevalence of COPD varies substantially by region and death rates attributed to COPD are twofold greater in South-West compared with North-East regions for reasons that are not fully understood.

Physical activity in terms of body movements, walking time and standing time has been shown to be reduced in patients with severe COPD. However, it is currently unknown at which clinical stage of the disease limitations of physical activity are first displayed. Furthermore, the relationships between physical activity and clinical characteristics reflecting the disease severity, such as the degree of airway obstruction, distance walked in 6 min, self-reported grade of dyspnea and clinical stages of COPD, need to be investigated as, to date, data are inconclusive or have never been evaluated. For example, some studies have found substantial correlations between airway obstruction and physical activity, while others found no or only loose relationships. Previous studies indicate that the 6-min walking distance (6MWD) might best reflect physical activity, while a recent study found airway obstruction to correlate with physical activity better than 6MWD.

ELIGIBILITY:
Inclusion criteria

1. Smokers and Non- Smokers.
2. Age between 18 to 60 years.
3. Both Male and Female

Exclusion criteria

1. Subjects with COPD Exacerbations
2. Subjects with respiratory complication others than CPOD
3. Bed bound subjects with CPOD

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Researcher will visit selected hospital setting with questionnaire and Consent form. Consent form will be signed from patient prior to questionnaire. IPAQ Questionnaire will be given and briefly elaborated before filling. 6MVT and spirometry measurements will be taken after and documented.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | Day 1
  IPAQ Urdu version will be used to document Physical Activity
6 minute Walk Test (6MWT) | Day 1
  6 Minute Walk Test is used to measure cardiovascular health
Forced Expiratory Volume 1 Sec | Day 1
  Forced Expiratory Volume 1 Sec is used to measure respiratory health
Forced vital capacity (FVC) | Day 1
  Forced vital capacity (FVC) is used to measure respiratory health
FEV1/FVC | Day 1
  FEV1/FVC ratio is used to measure respiratory health
Peak expiratory flow (PEF) | Day 1
  Peak expiratory flow (PEF) is used to measure respiratory health

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabiliation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bacharier LB, Beigelman A, Calatroni A, Jackson DJ, Gergen PJ, O'Connor GT, Kattan M, Wood RA, Sandel MT, Lynch SV, Fujimura KE, Fadrosh DW, Santee CA, Boushey H, Visness CM, Gern JE; NIAID sponsored Inner-City Asthma Consortium. Longitudinal Phenotypes of Respiratory Health in a High-Risk Urban Birth Cohort. Am J Respir Crit Care Med. 2019 Jan 1;199(1):71-82. doi: 10.1164/rccm.201801-0190OC. PMID 30079758
- [Background] Kurmi OP, Davis KJ, Hubert Lam KB, Guo Y, Vaucher J, Bennett D, Wang J, Bian Z, Du H, Li L, Clarke R, Chen Z. Patterns and management of chronic obstructive pulmonary disease in urban and rural China: a community-based survey of 25 000 adults across 10 regions. BMJ Open Respir Res. 2018 Feb 19;5(1):e000267. doi: 10.1136/bmjresp-2017-000267. eCollection 2018. PMID 29531747
- [Background] Aghilinejad M, Kabir-Mokamelkhah E, Nassiri-Kashani MH, Bahrami-Ahmadi A, Dehghani A. Assessment of Pulmonary Function Parameters and Respiratory Symptoms in Shipyard Workers of Asaluyeh City, Iran. Tanaffos. 2016;15(2):108-111. PMID 27904543
- [Background] Mesquita R, Spina G, Pitta F, Donaire-Gonzalez D, Deering BM, Patel MS, Mitchell KE, Alison J, van Gestel AJ, Zogg S, Gagnon P, Abascal-Bolado B, Vagaggini B, Garcia-Aymerich J, Jenkins SC, Romme EA, Kon SS, Albert PS, Waschki B, Shrikrishna D, Singh SJ, Hopkinson NS, Miedinger D, Benzo RP, Maltais F, Paggiaro P, McKeough ZJ, Polkey MI, Hill K, Man WD, Clarenbach CF, Hernandes NA, Savi D, Wootton S, Furlanetto KC, Cindy Ng LW, Vaes AW, Jenkins C, Eastwood PR, Jarreta D, Kirsten A, Brooks D, Hillman DR, Sant'Anna T, Meijer K, Durr S, Rutten EP, Kohler M, Probst VS, Tal-Singer R, Gil EG, den Brinker AC, Leuppi JD, Calverley PM, Smeenk FW, Costello RW, Gramm M, Goldstein R, Groenen MT, Magnussen H, Wouters EF, ZuWallack RL, Amft O, Watz H, Spruit MA. Physical activity patterns and clusters in 1001 patients with COPD. Chron Respir Dis. 2017 Aug;14(3):256-269. doi: 10.1177/1479972316687207. Epub 2017 Feb 24. PMID 28774199
- [Background] Rocha FR, Bruggemann AK, Francisco DS, Medeiros CS, Rosal D, Paulin E. Diaphragmatic mobility: relationship with lung function, respiratory muscle strength, dyspnea, and physical activity in daily life in patients with COPD. J Bras Pneumol. 2017 Jan-Feb;43(1):32-37. doi: 10.1590/S1806-37562016000000097. PMID 28380186